CLINICAL TRIAL: NCT01017133
Title: Assessing Hypoxia by 18F-EF5 PET Scanning and Glycolysis by 18FFDG PET Scanning in Subjects With Non-Small Cell Lung Cancer
Brief Title: Fluorine F18-EF5 and Fludeoxyglucose F18 Positron Emission Tomography in Assessing Hypoxia and Glycolysis in Patients With Stage I, Stage II, or Stage III Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UPCC 01509
Record Dates: First submitted 2009-11-18; First posted 2009-11-20 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Other): With 6 weeks prior to surgery, patients undergo fluorine F18 (18F)-EF5 PET at 10 minutes and 90 minutes after injection of 18F-EF5. Patients also undergo fludeoxyglucose F18 (18F-FDG) PET at 1 hour and 3 hours after injection of 18F-FDG.
  Interventions: Radiation: fludeoxyglucose F 18; Radiation: Fluorine F 18 EF5; Procedure: Positron emission tomography

INTERVENTIONS:
Radiation: fludeoxyglucose F 18 — Given IV
  Other Names: 18FDG, FDG, Fluorine-18 2-Fluoro-2-deoxy-D-Glucose, fluorodeoxyglucose F18
Radiation: Fluorine F 18 EF5 — Given IV
  Other Names: 18F-EF5
Procedure: Positron emission tomography — Undergo scan
  Other Names: FDG-PET, PET, PET scan, tomography, emission computed

SUMMARY:
RATIONALE: Diagnostic procedures, such as positron emission tomography, using the drug fluorine F18-EF5 to find oxygen and fludeoxyglucose F18 to find sugar in tumor cells may help in planning treatment for patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
PURPOSE: This clinical trial is studying fluorine F18-EF5 and fludeoxyglucose F18 positron emission tomography in assessing hypoxia and glycolysis in patients with stage I, stage II, or stage III non-small cell lung cancer.Detailed DescriptionOBJECTIVES:

I. To determine whether there is an association between Akt activation and hypoxia as determine by 18F-EF5 PET scanning in patients with NSCLC.

II. To determine whether there is an association between Akt activation and increased glycolysis as determined by 18F-FDG PET imaging in patients with NSCLC.

OUTLINE: Within 6 weeks prior to surgery, patients undergo fluorine F18 (18F)-EF5 PET at 10 minutes and 90 minutes after injection of 18F-EF5. Patients also undergo fludeoxyglucose F18 (18F-FDG) PET at 1 hour and 3 hours after injection of 18FFDG.

After completion of study treatment, patients are followed periodically for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a histologically confirmed NSCLC or clinical and imaging evidence of a de novo mass that is likely to be a NSCLC, stage I, II, or IIIA, for which surgery would be indicated for routine medical indications
* ECOG performance status between 0 and 2
* Subjects must sign an informed consent document that indicates they are aware of the investigational nature of the treatment in this protocol as well as the potential risks and benefits
* WBC > 2,000/mm^3
* Platelet count > 100,000/mm^3
* Total bilirubin
* Serum AST and ALT
* Serum creatinine
* Negative serum pregnancy test if a female of childbearing age

Exclusion Criteria:

* History of allergic reactions attributed to Flagyl (metronidazole), which has a chemical structure similar to EF5
* Uncontrolled intercurrent illness that would limit compliance with study requirements
* Pregnant women and women who are breastfeeding are excluded
* Subjects who have been treated with neoadjuvant radiation or chemotherapy prior to their biopsy or excision are excluded because the impact of these therapies upon the degree of hypoxia of the tumor is unknown

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2009-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
P-Akt in tumor cells as assessed by immunohistochemistry
Tumor hypoxia as assessed by 18F-EF5 PET imaging
Tumor Glycolysis as assessed by 18F-FDG PET imaging
Progression-free survival
Overall survival
Toxicity assessed by CTCAE v3.0

CONTACTS AND LOCATIONS:
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States